CLINICAL TRIAL: NCT05352906
Title: Accuracy of Handheld and Non-contact Tonometry in Clinical Practice
Brief Title: Accuracy of Handheld and Non-contact Tonometry
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Ahmed Abdelshafy, Lecturer of Ophthalmology, Benha University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: RC-10-2022
Record Dates: First submitted 2022-04-25; First posted 2022-04-29 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Glaucoma; Intraocular Pressure; Glaucoma, Suspect
Keywords: Glaucoma; Suspect; Tonometer; Air-puff
MeSH Terms: conditions — Glaucoma; Ocular Hypertension | interventions — Intraocular Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Contact goldman applanation tonometry (Active Comparator): The standard contact tonometer
  Interventions: Diagnostic Test: Intraocular pressure
- Handheld digital contact tonometer (Active Comparator): A contact digital tonometer's pen.
  Interventions: Diagnostic Test: Intraocular pressure
- Non-contact air-puff tonometer (Active Comparator): A non-contact tonometer based on air-puff and corneal hysteresis.
  Interventions: Diagnostic Test: Intraocular pressure

INTERVENTIONS:
Diagnostic Test: Intraocular pressure — Measurements of intraocular pressure in millimeter mercury (mmHg).

SUMMARY:
Monitoring the intraocular pressure (IOP) is one of the most important tests used in follow-up among glaucoma suspects and confirmed glaucomatous patients.

DETAILED DESCRIPTION:
In tertiary hospitals, IOP screening is an important tool to confirm glaucomatous eyes. Inaccurate measurements may lead to missed diagnosis or false positive results that may affect patients' quality of life.

There are many devices produced to measure IOP, the commonest one is Goldman contact tonometry, the aim of this study is to compare the results of new developed tonometers to the standard applanation tonometer.

ELIGIBILITY:
Inclusion Criteria:

* All subjects seeking regular check-up in glaucoma clinic at banha university hospital.
* Glaucoma suspects and glaucomatous patients that visit glaucoma clinic for regular IOP measurements.

Exclusion Criteria:

* Patients that will refuse to measure IOP again with other devices.
* patients with previous corneal surgeries or scar that may alter the measurements of the tonometer s (as previous keratoplasty, trauma or opacities).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2022-04-20 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-01-30 (Estimated)

PRIMARY OUTCOMES:
Accuracy of air-puff tonometry | Immediately after goldman applanation tonometry test for each eye.
  Comparing IOP measurements in (mmHg) between standard goldman applanation tonometry and air-puff non-contact tonometry.

SECONDARY OUTCOMES:
Accuracy of handheld tonometry | Immediately after goldman applanation tonometry test for each eye.
  Comparing IOP measurements in (mmHg) between standard goldman applanation tonometry and handheld contact tonometry.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed A Abdelshafy, MD, Principal Investigator — Benha University
Locations (1):
- Ahmed Abdelshafy, Banhā, QA, Egypt

IPD SHARING:
Plan to Share IPD: Undecided